CLINICAL TRIAL: NCT07187193
Title: Efficacy and Safety of Low-Dose Cytarabine Combined With Thalidomide in the Treatment of Adult Patients With Untreated Langerhans Cell Histiocytosis: A Prospective, Multicenter, Single-Arm Study.
Brief Title: Efficacy and Safety of Low-Dose Cytarabine Combined With Thalidomide in Adult Patients With Untreated LCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH006
Record Dates: First submitted 2025-08-25; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Cytarabine; Thalidomide

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, single-arm study.Planned enrollment of 50 patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newly diagnosed LCH patients (Experimental): (1) The histopathological diagnosis of LCH is confirmed; (2) Multi-system involvement or single-system with multiple lesions; (3) No prior systemic treatment (patients who have only received local radiotherapy or surgery are eligible);
  Interventions: Drug: Cytarabine (Ara-C); Drug: Thalidomide (100mg)

INTERVENTIONS:
Drug: Cytarabine (Ara-C) — The treatment regimen consists of Ara-C administered at a dose of 100 mg/m² from days 1 to 5, combined with thalidomide at a dose of 100 mg from days 1 to 35, repeated every 35 days for a total of 12 cycles. Following this, thalidomide will be given as monotherapy at a dose of 100 mg from days 1 to 28, administered every 28 days for an additional 12 cycles of maintenance treatment. In total, participants will undergo 24 cycles of treatment.
Drug: Thalidomide (100mg) — The treatment regimen consists of AraC administered at a dose of 100 mg/m² from days 1 to 5, combined with thalidomide at a dose of 100 mg from days 1 to 35, repeated every 35 days for a total of 12 cycles. Following this, thalidomide will be given as monotherapy at a dose of 100 mg from days 1 to 28, administered every 28 days for an additional 12 cycles of maintenance treatment. In total, participants will undergo 24 cycles of treatment.

SUMMARY:
Treatment of Adult Patients with Newly Diagnosed Langerhans Cell Histiocytosis (LCH) Using a Low-Dose Cytarabine Combined with Thalidomide Regimen.

DETAILED DESCRIPTION:
AraC 100 mg/m² d1-5+ thalidomide 100mg d1-35, q35 days ,for a total of 12 cycles;followed by thalidomide 100mg, qd1-28 q28d,for a total of 12 cycles of monotherapy maintenance reatment;

ELIGIBILITY:
Inclusion Criteria:

* Clearly diagnose and treat adult patients with multisystem or single-system multifocal LCH;
* Aged between 18 and 70 years;
* Multisystem involvement or single-system multifocal disease;
* No prior systemic treatment (patients who have only received local radiotherapy or surgery may be enrolled);
* ECOG performance status score ≤ 2;
* Judged by clinicians as suitable for treatment with this protocol;
* Patients or their families able to understand the study protocol and willing to participate in the study, providing written informed consent.

Exclusion Criteria:

* Patients with LCH involving the central nervous system;
* Single-system single-lesion LCH;
* Subjects who have undergone major surgery within 4 weeks prior to the first dose in the study;
* Subjects who have received radiotherapy within 4 weeks prior to the first dose in the study; subjects with a history of myocardial infarction within the past year;
* Patients with New York Heart Association (NYHA) class 3 or 4 congestive heart failure, or a history of NYHA class 3 or 4 congestive heart failure;
* Pregnant or lactating women;
* Abnormal liver and kidney function: creatinine level ≥176.8μmol/l (2mg/dl), transaminase and bilirubin levels more than 2 times the upper limit of normal (for LCH patients with liver involvement, bilirubin levels more than 10 times the upper limit of normal);
* Abnormal blood counts: absolute neutrophil count less than 1×10^9/L, platelet count less than 50×10^9/L;
* Patients or their families unable to understand the conditions and objectives of this study;
* Any other circumstances in which the investigator deems the patient unsuitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2027-04-12 (Estimated); Study Completion 2027-04-13 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | From enrollment to the end of treatment until 3 years
  The primary endpoint was event-free survival (EFS), with events defined as poor response (stable disease or progressive disease) to cytarabine and thalidomide therapy, or death from any cause. EFS was measured from initiation of cytarabine and thalidomide therapy until the date of the first documented event, with censoring of patients without events at the last follow-up.

SECONDARY OUTCOMES:
Overall survival (OS) | From enrollment to the end of treatment until 3 years
  OS was defined as the time from cytarabine and thalidomide initiation to death or last follow-up.
Overall response rate (ORR) | From enrollment to the end of treatment until 3 years
  The overall response rate (ORR) was defined as the cumulative proportion of patients achieving either a complete response (CR) or partial response (PR) following therapy.
Adverse events | From enrollment to the end of treatment until 3 year
  Toxicities were recorded and graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

OTHER OUTCOMES:
FACT-G (Functional Assessment of Cancer Therapy-General) | From enrollment to the end of treatment until 3 years
  Score of FACT-G (Functional Assessment of Cancer Therapy-General)
Correlation between next-generation sequence (NGS) / circulating free DNA (cfDNA) and efficacy/EFS | From enrollment to the end of treatment until 3 years
  Correlation between the positivity of next-generation sequence (NGS) / circulating free DNA (cfDNA) and efficacy/EFS

CONTACTS AND LOCATIONS:
Overall Officials: Xinxin XX Cao, doctor, Study Chair — NCC, CICAMS
Locations (1):
- Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No